CLINICAL TRIAL: NCT01959607
Title: A Single-center, Open-label, Randomized, Controlled, Crossover Study to Investigate the Nicotine Pharmacokinetic Profile and Safety of THS 2.2 Following Single Use in Healthy Smokers Compared to Conventional Cigarettes and Nicotine Gum
Brief Title: Nicotine Pharmacokinetic Profile and Safety of the Tobacco Heating System 2.2 (THS 2.2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZRHR-PK-02-JP; ZRHR-PK-02-JP (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Smoking
Keywords: Smoking; Nicotine absorption; Candidate modified risk tobacco product; Cigarettes; Nicotine Replacement Therapy gum (NRT gum)
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- THS 2.2 then CC (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of THS 2.2)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of CC).
  Interventions: Other: THS 2.2; Other: CC
- CC then THS 2.2 (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of CC)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of THS 2.2).
  Interventions: Other: THS 2.2; Other: CC
- THS 2.2 then NRT (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of THS 2.2)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single administration of NRT gum [Nicorette® 2mg]).
  Interventions: Other: THS 2.2; Other: NRT Gum
- NRT then THS 2.2 (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single administration of NRT gum [Nicorette® 2mg])
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of THS 2.2).
  Interventions: Other: THS 2.2; Other: NRT Gum

INTERVENTIONS:
Other: THS 2.2 — Single use of the Tobacco Heating System 2.2 (THS 2.2)
Other: CC — Single use of subject's own cigarette (CC)
  Arms: CC then THS 2.2; THS 2.2 then CC
Other: NRT Gum — Single administration of the nicotine replacement therapy (NRT) 2 mg gum (Nicorette® 2mg)
  Arms: NRT then THS 2.2; THS 2.2 then NRT

SUMMARY:
The overall goal of the study is to evaluate the pharmacokinetic (PK) profile (rate and the amount of nicotine absorbed) following a single use of the THS 2.2, a candidate Modified Risk Tobacco Product, compared to the PK profiles from a single use of a cigarette (CC) and from a single use of nicotine gum in a Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese.
* Smoking, healthy subject as judged by the Investigator.
* Subject smokes at least 10 commercially available CCs per day (no brand restrictions) for the last 4 weeks.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of a drug (whichever is longer) which has an impact on CYP2A6 activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masayuki Sugimoto, MD PhD, Principal Investigator — Koganeibashi Sakura Clinic; Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (1):
- Koganeibashi Sakura Clinic, 2-11-25, Sakuracho, Koganei-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 31 July 2013
  At admission (Day -1), all the subjects performed a product trial (Tobacco Sticks and subsequently NRT gum).
  From enrollment, they were asked to remain abstinent from smoking for at least 24 hours (Day 0) before being randomized on Day 1 into one of four product use sequences.
Pre-assignment Details: Enrolled population = 65 subjects: 3 subjects exposed to THS 2.2 and NRT gum at Admission but not randomized and 62 randomized to one of the four product use sequences described below:
  * Product Use Sequence "THS 2.2 then CC": 22 subjects
  * Product Use Sequence "CC then THS 2.2": 22 subjects
  * Product Use Sequence "THS 2.2 then NRT": 9 subjects
  * Product Use Sequence "NRT then THS 2.2": 9 subjects
Groups:
- THS 2.2 Then NRT: Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of THS 2.2)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single administration of NRT gum [Nicorette ® 2mg]).
- NRT Then THS 2.2: Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single administration of NRT gum [Nicorette ® 2mg])
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of THS 2.2).
Period: Washout Period of 24 Hrs. (Day 0)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NRT | NRT Then THS 2.2
Started | 22 | 22 | 9 | 9
Completed | 22 | 22 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: First Intervention (Day 1)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NRT | NRT Then THS 2.2
Started | 22 | 22 | 9 | 9
Completed | 21 | 21 | 9 | 9
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: Washout Period of 24 Hrs. (Day 2)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NRT | NRT Then THS 2.2
Started | 21 | 21 | 9 | 9
Completed | 21 | 21 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (Day 3)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NRT | NRT Then THS 2.2
Started | 21 | 21 | 9 | 9
Completed | 21 | 21 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of 65 subjects:
  * 62 subjects randomized to one of four product use sequences
  * three subjects exposed to THS 2.2 and NRT gum during the product trial on Day -1 but not randomized.
Groups:
- THS 2.2 - CC: This population was randomized to the following product use sequence:
  "THS 2.2 then CC"
- CC -THS 2.2: This population was randomized to the following product use sequence:
  "CC then THS 2.2"
- THS 2.2 - NRT: This population was randomized to the following product use sequence:
  "THS 2.2 then NRT"
- NRT - THS 2.2: This population was randomized to the following product use sequence:
  "NRT then THS 2.2"
- Enrolled But Not Randomized: This population comprised enrolled subjects who tried the THS 2.2 at Admission (Day -1) but were not randomized to a product use sequence.
- Total: Total of all reporting groups
Arm/Group | THS 2.2 - CC | CC -THS 2.2 | THS 2.2 - NRT | NRT - THS 2.2 | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 22 | 22 | 9 | 9 | 3 | 65
Age, Customized [Mean (Standard Deviation); unit: years]
  Between 23 and 65 years | 32.9 (7.56) | 32.7 (9.84) | 34.7 (12.36) | 36.9 (8.71) | 42.7 (11.85) | 34.1 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 6 | 4 | 0 | 34
  Male | 11 | 9 | 3 | 5 | 3 | 31
International Organization for Standardization (ISO) nicotine level [Number; unit: participants]
  ≤ 0.6 mg | 14 | 8 | 6 | 4 | 0 | 32
  > 0.6 to ≤ 1 mg | 8 | 14 | 3 | 5 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of THS 2.2, CC and NRT
Description: T0 = start of single product use.
  Derived from multiple blood sampling on Day 1 and Day 3 (1 blood sampling pre-product use and multiple blood sampling over 24 hours post-product use).
  Geometric Least Squares means are provided.
Time Frame: Blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0
Population: PK populations consisted of all the randomized subjects who completed at least 1 of the single use days (Days 1 or 3), and for whom at least 1 PK parameter could be derived. Subjects with major protocol deviations that impacted the evaluability of the results were excluded from the PK populations.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- THS 2.2 - Group 1; CC - Group 1: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "THS 2.2 then CC"
  * Sequence "CC then THS 2.2"
- THS 2.2 - Group 2; NRT - Group 2: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "THS 2.2 then NRT"
  * Sequence "NRT then THS 2.2"
Arm/Group | THS 2.2 - Group 1 | CC - Group 1 | THS 2.2 - Group 2 | NRT - Group 2
Number analyzed (Participants) | 42 | 42 | 18 | 18
ng/mL | 14.30 [12.43 to 16.45] | 13.82 [12.01 to 15.89] | 11.53 [7.49 to 17.74] | 4.80 [3.11 to 7.39]
Statistical Analysis 1: Comparison: THS 2.2 - Group 1 vs CC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of THS 2.2:CC) for Cmax, therefore, there was no statistical hypothesis to be tested for this objective; Test type: Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 103.50, 95% CI 2-sided [84.94 to 126.11] — LS mean ratio (THS 2.2 - Group 1:CC - Group 1)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (Pre-product Use) to Last Time Point [AUC(0-last)] Following Single Use of THS 2.2, CC and NRT
Description: as for outcome 1
Time Frame: Blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | THS 2.2 - Group 1 | CC - Group 1 | THS 2.2 - Group 2 | NRT - Group 2
Number analyzed (Participants) | 42 | 42 | 18 | 18
ng*h/mL | 23.75 [21.76 to 25.94] | 24.66 [22.58 to 26.92] | 18.92 [13.30 to 26.91] | 14.88 [10.46 to 21.17]
Statistical Analysis 1: Comparison: THS 2.2 - Group 1 vs CC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of THS 2.2:CC) for AUC(0-last), therefore, there was no statistical hypothesis to be tested for this objective; Test type: Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 96.34, 95% CI 2-sided [85.10 to 109.07] — LS mean ratio (THS 2.2 - Group 1:CC - Group 1)

ADVERSE EVENTS:
Time Frame: From informed consent form (ICF) signature until the end of the safety follow-up period (7 days after discharge of the subject)
Description: The safety population consisted of 65 subjects (62 randomized subjects and 3 subjects exposed to THS 2.2 and NRT gum during the product trial on Day -1 but not randomized). Adverse events were reported according to the product use sequence and intervention. Adverse events by intervention are reported here.
Groups:
- THS 2.2 Use: This population used THS 2.2 as part of their randomized product use sequence
- CC Use: This population used CC as part of their randomized product use sequence
- NRT Gum Use: This population used NRT Gum as part of their randomized product use sequence
Arm/Group | THS 2.2 Use | CC Use | NRT Gum Use | Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/18 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/18 | 0/3
Other Adverse Events (participants affected / at risk) | 1/44 | 1/44 | 2/18 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Use (N=44) | CC Use (N=44) | NRT Gum Use (N=18) | Enrolled But Not Randomized (N=3)
Dysphoria (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2013-06-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT01959607/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT01959607/SAP_001.pdf